CLINICAL TRIAL: NCT00363467
Title: A Pilot Study of Intravenous, Targeted-Dose Busulfan Monotherapy as Conditioning for Autologous Hematopoietic Progenitor Cell Transplantation in High-Risk AML
Brief Title: Busulfan Monotherapy as Conditioning for Autologous Hematopoietic Progenitor Cell Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: ESP Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MCC-14604
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2011-09-30 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2011-08

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Busulfan; Acute myeloid leukemia (AML); Hematopoietic Stem Cell Transplantation (HSCT); Dendritic cells; Bone marrow transplantation; PBSC mobilization; Autologous stem cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Leukapheresis; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Hematopoietic Progenitor Cell Transplantation (Other): G-CSF Mobilization Leukepheresis Busulfan Stem Cell Reinfusion
  Interventions: Drug: G-CSF; Drug: Leukapheresis; Drug: Busulfan; Procedure: Stem cell reinfusion

INTERVENTIONS:
Drug: G-CSF — Mobilization Option 1:Twenty-four to 48 hours following completion of consolidation chemotherapy, patients will begin to receive G-CSF at 10 mcg/kg twice daily subcutaneously.
  Mobilization Option 2: If patients have recovered hematologically from consolidation chemotherapy, they may receive G-CSF at 10 mcg/kg twice daily subcutaneously.
  Other Names: filgrastim or NeupogenR
Drug: Leukapheresis — leukapheresis
Drug: Busulfan — Busulfan IV daily x 4 days (transplantation days -5,-4,-3,-2). The day -5 and -4 dose will be 130mg/m2
  Other Names: Busulfan (MyleranR, Busulfex™)
Procedure: Stem cell reinfusion — autologous stem cell transplant

SUMMARY:
During the pre-transplantation phase (following completion of consolidation chemotherapy), patients will begin to receive G-CSF at 10 mcg/kg twice daily; leukapheresis will also be given until a target goal for recipient body weight is obtained, or up to a maximum of 5 days. Conditioning/Preparative therapy will follow PBSC collection for up to 30 days with Busulfan IV daily x 4 days; subsequent doses will be adjusted based on pharmacokinetic (plasma level)monitoring. Following 1 day of rest, stem cell reinfusion will begin with supportive care. During follow-up, patients will be monitored out to 730 days.

DETAILED DESCRIPTION:
1. Pre- Transplantation Phase -

   1. Twenty-four to 48 hours following completion of consolidation chemotherapy, patients will begin to receive G-CSF at 10 mcg/kg twice daily subcutaneously. Alternatively, patients may receive G-CSF alone (same dose) as mobilization therapy.
   2. Leukapheresis will begin day 4 of G-CSF administration and proceed according to institutional guidelines. Leukapheresis will continue until a target goal for recipient body weight is obtained, or up to a maximum of 5 days. A minimum recipient body weight is required to proceed to transplantation.
2. Transplantation Phase

   a. Conditioning/Preparative therapy - up to 30 days following PBSC collection, patients will begin conditioning therapy with Busulfan IV daily x 4 days (transplantation days -5,-4,-3,-2). The day -5 and -4 dose will be 130mg/m2; subsequent doses will be adjusted based on pharmacokinetic monitoring.
   * Busulfan plasma level monitoring, collected around the first dose of busulfan b. Stem cell reinfusion - following 1 day of rest, previously collected autologous peripheral blood stem cells will be infused.
   * The administration of supportive measures (e.g. intravenous fluids, antihistamines) during stem cell reinfusion will be performed according to institutional guidelines.
3. Supportive care

   1. Antibiotic prophylaxis- according to hospital/institutional guidelines, and at the discretion of the treating physician.
   2. Growth factor support
   3. Transfusion support
   4. Prophylaxis for busulfan-induced seizures
4. During follow-up, patients will be seen at least weekly for the first month and there after periodically out to 730 days posttransplant. The following medical procedures will be done:

   * Medical history and physical exam (including concurrent meds, vital signs, performance status and weight)
   * Standard labs
   * Bone marrow aspirate and biopsy

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologically confirmed diagnosis of AML, in 1st complete remission, by a pathologic review at the H. Lee Moffitt Cancer Center and Research Institute. Any induction/consolidation regimen is permitted.
* General Inclusion Criteria:

  1. Age 56-74
  2. Able to give informed consent
  3. Hepatic and renal function: normal bilirubin, AST and ALT less than or equal to 2x normal limits, serum creatinine less than or equal to 1.5x normal
  4. Left ventricular ejection fraction (LVEF) must be in normal range
  5. FEV1 AND DLCO greater than or equal to 50% predicted (at planned time of transplantation)
  6. ECOG PS less than or equal to 2 (at planned time of transplantation)
* Disease Specific Inclusion Criteria:

  1. Adverse-risk karyotype (del 5/5q, 7/7q, 3q, greater than or equal to 3 abnormalities):
  2. Intermediate-risk karyotype [46 XY, +8, -Y, +6, or any other isolated (<3 total) non-random abnormality not included in the adverse-risk category or favorable-risk category below]
* AML arising from antecedent hematologic disorder (e.g. MDS)
* Secondary AML (t-AML)

Exclusion Criteria:

* Acute Promyelocytic Leukemia(FAB M3) subtype
* Presence of (8;21) translocation or inversion 16/t(16;16) cytogenetic phenotype (i.e. favorable-risk AML)
* Eligible for and willing to undergo matched-sibling allogeneic transplantation
* Greater than 2 induction regimens required to achieve complete remission
* Duration of > 8 weeks between completion of induction chemotherapy and initiation of consolidation chemotherapy
* No prior malignancy is allowed, except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least 5 years.
* Prior extensive radiation therapy (>25% of bone marrow reserve)
* Concomitant radiation therapy, chemotherapy, or immunotherapy
* Intrinsic impaired organ function (as stated above)
* Active infection
* Positive serum pregnancy test in women who have not yet reached menopause (no menstrual periods for >12 months or who have not undergone tubal ligation or complete hysterectomy.
* Women who are breast-feeding
* Positive HIV testing
* Presence of CNS leukemia
* Uncontrolled insulin-dependent diabetes mellitus or uncompensated major thyroid or adrenal gland dysfunction
* Physical or psychiatric conditions that in the estimation of the PI or his designee place the patient at high-risk of toxicity or non-compliance

Ages: 56 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E Lancet, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffiitt Cancer Center Clinical Trials Website — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period May 15, 2006 through May 20, 2009; H. Lee Moffitt Cancer Center.
Pre-assignment Details: The study did not involve a wash-out period or group assignment.
Period: Overall Study
Arm/Group | Autologous Hematopoietic Progenitor Cell Transplantation
Started | 3
Completed | 2
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Autologous Hematopoietic Progenitor Cell Transplantation
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (2.828427)
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: 100-day Non-relapse Mortality
Description: 100-day non-relapse mortality is the number of participants who died before day 100 posttransplant from causes other than relapsed disease
Time Frame: 100 days post transplant
Population: Analysis was "per protocol"
Measure: Number; unit: participants
Arm/Group | Autologous Hematopoietic Progenitor Cell Transplantation
Number analyzed (Participants) | 2
participants | 0

2. Secondary Outcome: Successful Autologous Stem Cell Collection
Description: Number of subjects who were able to collect at least 2 million CD34+ cells/kg
Time Frame: At time of stem cell collection
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Autologous Hematopoietic Progenitor Cell Transplantation
Number analyzed (Participants) | 2
participants | 2

3. Secondary Outcome: Severe Regimen-related Toxicity
Description: Number of participants with severe regimen-related toxicity within 2 years posttransplant. Severe regimen-related toxicity was defined as CTC (version 3)grade 4.
Time Frame: up to 100 days post translant
Measure: Number; unit: participants
Arm/Group | Autologous Hematopoietic Progenitor Cell Transplantation
Number analyzed (Participants) | 2
participants | 2

4. Secondary Outcome: 1 Year Event-free Survival
Description: Number of participants alive and without disease relapse at 1 year posttransplant
Time Frame: 1 year post transplant
Measure: Number; unit: participants
Arm/Group | Autologous Hematopoietic Progenitor Cell Transplantation
Number analyzed (Participants) | 2
participants | 2

5. Secondary Outcome: 1 Year Overall Survival
Description: Number of participants alive at 1 year posttransplant
Time Frame: 1 year post transplant
Measure: Number; unit: participants
Arm/Group | Autologous Hematopoietic Progenitor Cell Transplantation
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Arm/Group | Autologous Hematopoietic Progenitor Cell Transplantation
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Two patients enrolled and transplanted out of 24 targeted transplant accrual goal. Due to poor enrollment study closed and no further analyses were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes